CLINICAL TRIAL: NCT05998083
Title: Investigation of the Effect of Purposeful Balance and Coordination Exercises on Attention and Quality of Life in Children Diagnosed With Special Learning Disabilities.
Brief Title: The Effectiveness of Purposeful Exercises in Children Diagnosed With Special Learning Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar71
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Lack of; Attention, With Hyperactivity (ADHD); Specific Learning Disability
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: In addition to the individual training program they received from the special training center, the experimental group was given goal-oriented balance and coordination exercises for 40 minutes, 2 days a week.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): continued their normal education and physiotherapy
  Interventions: Other: control
- experimental group (Experimental): they continued their normal training and physiotherapy, in addition, purposeful balance and coordination exercises were given for 40 minutes a day, 2 days a week for 8 weeks.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — In addition to the individual support training program, the exercise group was given a balance and coordination exercise protocol including 40 minutes, 2 days a week.
  These exercises are:
  It consisted of warm-up (10 minutes), purposeful balance and coordination exercises (20 minutes), and cool-down (10 minutes) exercises.
  Balance and coordination exercises with purpose were created with a series of exercises based on copying the shape of the blocks on the cards placed at the beginning of a track consisting of stations at the end of the track. The stations were composed of "hopscotch station", "tandem walking station in one line", "bounce station", "bucketing ping pong balls station" and "eight running stations".
  Arms: experimental group
Other: control — The control group continued only the individual support education program.
  Arms: control group

SUMMARY:
The aim of the study is to examine the effect of purposeful balance and coordination exercises on attention and quality of life in children diagnosed with special learning disabilities.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled trial, and children aged 7-17 who were diagnosed with "Special Learning Disability" in a special education center in Kocaeli-Darica were included as a sample. Children were divided into experimental and control groups by randomization. In addition to the individual training program they received from the special training center, the experimental group was given goal-oriented balance and coordination exercises for 8 weeks, 2 days a week for 40 minutes. The control group continued only the individual training program. All participants and their parents were informed about the study, and an informed consent form was obtained from the participants and their parents. In order to collect data from the participants; "Leisure Time Activity Questionnaire for Children" to determine physical activity levels, "Quality of Life Assessment Questionnaire for Children" to determine their quality of life, "Bruininks-Oseretsky Motor Proficiency Test 2 short form" to evaluate motor skills, "Burdon Attention Test" to measure attention level used. These tests and forms were repeated before starting the study and at the end of the study. Pre- and post-intervention data were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Special Learning Disabilities
* To be between the ages of 7-15
* To attend the special education and rehabilitation center and individual support training program regularly.
* Not having exercise intolerance or any disease that prevents exercise
* The child's willingness to participate in the study and the consent of the parent to participate in the study

Exclusion Criteria:

* Having physical or psychological disorders in addition to the diagnosis of Special Learning Disabilities (ADHD, etc.)
* Being diagnosed with Special Learning Disabilities and not complying with the age range
* Not attending the individual training program regularly
* Parents not giving consent for the child to participate in the study

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
The Quality of Life Scale for Children (QoL-C) | 10 weeks
  Quality of Life Scale for Children, parent form for children or adolescents 2-4, 5-7, 8-12, 13-18 years old, and self for children or adolescents 5-7, 8-12, 13-18 years old It consists of a total of 7 forms, including a notification form. This scale questions the last month of children and adolescents. It was developed as a Likert-type scale with 3 options for children aged 5-7 and 5 options for children and adolescents aged 8-18. Items are scored between 0-100. The answer to the question is scored 100 if it is marked as never, 75 if it is marked as rarely, 50 if it is marked as sometimes, 25 if it is marked as often, and 0 if it is marked as almost always. The total score is obtained by summing the scores and dividing by the number of items filled. The score obtained is directly proportional to the quality of life.
Leisure Activity Questionnaire for Children (CPAQ) | 10 weeks
  The form was filled by the children and their exercise levels were determined by calculations. MET values were classified as low, medium, high and moderately high. Low-intensity activities of 3 METs or less per hour are moderate and high-intensity activities of 3 METs and above. It is considered as moderate (3-5.9 MET), high intensity (6 MET and above), and medium-high intensity (3 MET and above).
bourdon attention test | 10 weeks
  Bourdon Test (also dubbed a/b/q Test, ABQ) is an approach to measure focus and attentiveness that requires its taker to spot and cross out the query chars a, b and q in a potpourri of letters.
  The test consists of two forms. The first is to find and mark certain letters among mixed book letters; the second one is in the form of finding and marking certain figures among the figures given as mixed. There are a total of 660 letters in the letter form of the test. In the letter form, certain letters are required to be found among the letters. There is no template created, and the practitioner can choose the letters or shapes he wants and ask the children to mark them, so that the practitioner can create his own template.
bruninks oserertsky engine proficiency test-2(BOT-2) | 10 weeks
  BOT-2 measures fine and gross motor proficiency, with subtests that focus on stability, mobility, strength, coordination, and object manipulation. The test is tailored to school-aged children and young adults among the ages of 4-21 years, who have varying motor control abilities ranging from normal to mild or moderate.In both the BOT-2 short form (SF) this scale is used to transform the standard score to final categories (1 - well below average; 2 - below average; 3 - average; 4 - above average; 5 - well above average).The four motor-area composite standard scores, discussed below, range from 27 on Manual Coordination to 61 on Fine Manual Control.

CONTACTS AND LOCATIONS:
Overall Officials: Elif PUNAR, Study Chair — Uskudar University; Turgay ALTUNALAN, Study Chair — Karadeniz Technical University
Locations (1):
- Özel Eğitim Merkezi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanchet M, Assaiante C. Specific Learning Disorder in Children and Adolescents, a Scoping Review on Motor Impairments and Their Potential Impacts. Children (Basel). 2022 Jun 15;9(6):892. doi: 10.3390/children9060892. PMID 35740829
- [Background] Hallawell B, Stephens J, Charnock D. Physical activity and learning disability. Br J Nurs. 2012 May 24-Jun 13;21(10):609-12. doi: 10.12968/bjon.2012.21.10.609. PMID 22875298
- [Background] Bluechardt MH, Wiener J, Shephard RJ. Exercise programmes in the treatment of children with learning disabilities. Sports Med. 1995 Jan;19(1):55-72. doi: 10.2165/00007256-199519010-00005. PMID 7740247
- [Background] Fathi Azar E, Mirzaie H, Jamshidian E, Hojati E. Effectiveness of perceptual-motor exercises and physical activity on the cognitive, motor, and academic skills of children with learning disorders: A systematic review. Child Care Health Dev. 2023 Nov;49(6):1006-1018. doi: 10.1111/cch.13111. Epub 2023 Mar 7. PMID 36872844
- [Background] Maiano C, Hue O, Morin AJS, Lepage G, Tracey D, Moullec G. Exercise interventions to improve balance for young people with intellectual disabilities: a systematic review and meta-analysis. Dev Med Child Neurol. 2019 Apr;61(4):406-418. doi: 10.1111/dmcn.14023. Epub 2018 Sep 19. PMID 30230530
- [Derived] Punar E, Sevgin O. Effect of goal-directed perceptual-motor exercise on children with specific learning difficulties: a randomized controlled trial. BMC Pediatr. 2024 Dec 19;24(1):820. doi: 10.1186/s12887-024-05309-6. PMID 39695424